CLINICAL TRIAL: NCT06910215
Title: The Effectiveness of Elastic Therapeutic Taping in Pain Management After Sternotomy: A Randomized Controlled Double-Blind Study in Patients Undergoing Coronary Artery Bypass Grafting Surgery
Brief Title: Effect of Elastic Therapeutic Taping on Post-Sternotomy Pain in Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Alp Ozel, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIBU-FTR-AO-03
Record Dates: First submitted 2025-03-25; First posted 2025-04-04 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain; Sternotomy; Pain Management; Coronary Artery Bypass
Keywords: Postoperative Pain; Sternotomy; Kinesio Tape; Anxiety; Sleep Quality; Coronary Artery Bypass
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Elastic Therapeutic Taping Group (Experimental): Participants in this group will receive elastic therapeutic taping (kinesio taping) applied bilaterally 3 cm lateral to the sternotomy incision site. The tape will be applied with standardized tension and technique by a trained physiotherapist within 24 hours post-CABG surgery. The tape will remain in place for 48 hours. The goal is to assess the therapeutic effect of kinesio taping on postoperative pain and related outcomes.
  Interventions: Other: Elastic therapeutic taping
- Placebo Taping Group (Placebo Comparator): Participants in this group will receive placebo taping to the same area (3 cm lateral to the sternotomy incision), using the same type of tape but without any tension or therapeutic intent. The tape will be applied by the same trained team, in an identical manner visually, but with no mechanical stretch. The tape will also remain in place for 48 hours. This will help control for the placebo effect of the taping procedure.
  Interventions: Other: Placebo Elastic Therapeutic Taping
- Psychosocial Support Group (Sham Comparator): Participants in this group will receive elastic therapeutic tape applied to unrelated regions of the body (e.g., shoulder, back, or intercostal muscles) not associated with the surgical area. The purpose is to account for contextual or psychosocial effects of receiving an intervention. The tape will be applied without therapeutic intent for the surgical pain, and will stay in place for 48 hours.
  Interventions: Other: Therapeutic Taping on Non-Surgical Areas

INTERVENTIONS:
Other: Elastic therapeutic taping — Elastic therapeutic taping is a non-invasive method that uses a specially designed elastic cotton tape applied directly to the skin. In this study, it is used to support pain management after open-heart surgery (CABG via sternotomy). The tape is applied near the surgical site to gently lift the skin, which may help reduce pain, improve circulation, and support healing. The application is done by a trained physiotherapist following a standardized taping protocol. The tape remains on the skin for up to 48 hours.
  Arms: Elastic Therapeutic Taping Group
Other: Placebo Elastic Therapeutic Taping — In this group, the same type of elastic tape used in the therapeutic group is applied to the skin near the surgical area, but without any stretch or therapeutic technique. The tape does not provide physical support or intended therapeutic effects. It is used to help researchers understand whether any improvements are due to the taping itself or simply from receiving an intervention. The tape remains in place for up to 48 hours and is applied by trained personnel using a standardized, non-therapeutic method.
  Arms: Placebo Taping Group
Other: Therapeutic Taping on Non-Surgical Areas — In this group, elastic therapeutic tape is applied to body areas not directly related to the surgery, such as the shoulder, back, or rib area. The purpose is not to treat pain at the surgical site, but to simulate the experience of receiving a physical intervention. This approach helps researchers understand the potential impact of attention, expectation, or psychological support related to being part of a study. The tape is applied gently without therapeutic intent and stays on for up to 48 hours
  Arms: Psychosocial Support Group

SUMMARY:
This research study aims to find out whether elastic therapeutic taping can help reduce pain after heart surgery, specifically coronary artery bypass grafting (CABG), which is done using a surgical cut through the breastbone (sternotomy). This type of surgery often causes pain that makes it hard for patients to breathe deeply, move around, or recover quickly. Managing this pain in a safe and effective way is important for better healing and quality of life.

Elastic therapeutic taping is a method where special stretchy tape is applied to the skin to reduce pain and support the muscles. It is already used for other conditions like back or shoulder pain. In this study, researchers want to see if this taping method can also help people recover better after heart surgery by lowering pain, helping movement, and improving sleep and emotional well-being.

A total of 195 participants who had planned (elective) CABG surgery will be included in the study. People will be placed into one of three groups:

One group will get real elastic tape applied near the surgical area.

One group will get fake (placebo) tape that looks the same but has no medical effect.

One group will get a different kind of supportive treatment in other body areas.

Neither the patients nor the people measuring the results will know which group each person is in. This is called a "double-blind randomized controlled trial," which is the best way to get reliable results.

The researchers will check each participant's pain levels using a visual scale, and will also look at other things like oxygen levels, sleep quality, anxiety, how well they move, and how much pain medicine they use. These checks will happen several times in the first two days after surgery.

The taping is safe and non-invasive. Some people may experience mild skin irritation, but no serious side effects are expected. Participation is voluntary, and people can leave the study at any time. No payments will be made to participants, and all medical services related to the study will be free of charge.

This study is supported by Bolu Abant Izzet Baysal University. The results may help offer a new, drug-free option for managing pain after heart surgery and may improve patients' recovery experience.

DETAILED DESCRIPTION:
This randomized, controlled, double-blind clinical trial is designed to assess the efficacy of elastic therapeutic taping in reducing post-sternotomy pain in patients undergoing elective coronary artery bypass grafting (CABG) via median sternotomy. The study will be conducted at a single tertiary care center and will enroll 195 participants aged 18-75 years.

Participants will be randomized into three equal groups (n = 65 per group) using a computer-generated block randomization method. Allocation concealment will be maintained using sealed opaque envelopes. The interventions will be applied within 6-8 hours after extubation in the intensive care unit, and participants will be followed for 48 hours post-intervention.

Intervention Details:

Elastic Therapeutic Taping Group: Kinesio tape will be applied bilaterally, approximately 3 cm lateral to the sternotomy incision. The tape will be applied using standardized protocols with 25-35% stretch, following the muscle facilitation technique for pain relief and proprioceptive input.

Placebo Taping Group: Identical tape will be applied in the same locations, but without any stretch, and without following therapeutic taping principles. This group controls for the tactile and visual stimulus of taping.

Sham Taping (Contextual Support) Group: Tape will be applied to non-surgical, compensatory areas (e.g., shoulders, paravertebral region, or intercostal muscles) using a standard method, but in locations unrelated to the surgical site. This group is intended to control for the psychological and contextual effects of physical touch and therapist interaction.

All taping procedures will be performed by certified kinesio taping practitioners. The tape will remain in place for 48 hours unless early removal is required due to adverse skin reactions.

Blinding:

The study employs a double-blind design. Participants, outcome assessors, and data analysts will be blinded to group allocation. Intervention providers will not be involved in outcome assessment or data analysis.

Data Collection and Monitoring:

Primary and secondary outcome data will be collected at baseline (prior to intervention), and at 12, 24, and 48 hours post-intervention. Adherence to the intervention and any adverse events (e.g., skin irritation, allergic reaction) will be recorded. A dedicated safety officer will monitor for protocol adherence and unexpected complications.

Statistical Plan:

All analyses will follow an intention-to-treat approach. Descriptive statistics will summarize baseline characteristics. Normality will be assessed using the Shapiro-Wilk test. Between-group differences at each time point will be analyzed using one-way ANOVA or Kruskal-Wallis test. Repeated measures ANOVA or Friedman test will be used for within-group temporal comparisons. Bonferroni correction will adjust for multiple comparisons. Effect sizes (Cohen's d, partial eta squared) will be calculated.

Ethical Considerations:

The study protocol has been approved by the relevant institutional ethics committee. Written informed consent will be obtained from all participants. No experimental drugs or devices will be used. The tape used is CE-certified for medical use. The study adheres to the principles of the Declaration of Helsinki and Good Clinical Practice guidelines.

This study aims to provide high-quality evidence on the effectiveness of elastic therapeutic taping as a non-pharmacological intervention for managing early postoperative pain and improving recovery outcomes in CABG patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Undergoing elective coronary artery bypass graft (CABG) surgery via sternotomy
* Able to understand and communicate effectively
* Willing to provide informed consent

Exclusion Criteria:

* Presence of dermatological conditions or open wounds in the sternotomy area
* History of allergy to elastic therapeutic tape or adhesive materials
* Diagnosis of neurological or psychiatric conditions that may affect pain perception
* Currently taking medications that significantly alter pain sensitivity (e.g., neuropathic pain medications)
* Participation in another interventional clinical study within the past 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2025-12-24 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (Visual Analog Scale - VAS) | Baseline, 12 hours, 24 hours, and 48 hours after intervention
  Change in pain intensity will be assessed using the Visual Analog Scale (VAS), a 100 mm horizontal line where participants rate their pain from 0 (no pain) to 100 (worst imaginable pain).

SECONDARY OUTCOMES:
Oxygen Saturation (SpO₂) | Baseline, 12 hours, 24 hours, and 48 hours after intervention
  Peripheral oxygen saturation measured using a pulse oximeter to assess potential respiratory improvement.
Sleep Quality (VAS) | Baseline, 24 hours, and 48 hours after intervention
  Participants will rate their sleep quality using a Visual Analog Scale (0 = very poor, 100 = excellent).
Anxiety Level (VAS) | Baseline, 12 hours, 24 hours, and 48 hours post-intervention
  Participants will rate their anxiety level using a Visual Analog Scale (0 = no anxiety, 100 = extreme anxiety).
Functional Mobility (Timed Up and Go Test) | Baseline, 12 hours, 24 hours, and 48 hours after intervention
  Time (in seconds) taken by participants to rise from a chair, walk 3 meters, turn around, walk back, and sit down.
Analgesic Use | 0-48 hours post-intervention
  Total dosage of analgesic medication used during the first 48 hours post-surgery.
Length of Hospital Stay | From the date of surgery until hospital discharge, assessed up to 30 days postoperatively.
  Number of days from the date of surgery to the date of hospital discharge, as documented in the patient's medical record.
Fatigue Severity (VAS) | Baseline,12 hours, 24 hours, and 48 hours post-intervention
  Participants will rate their level of fatigue on a 100 mm Visual Analog Scale, where 0 indicates "no fatigue" and 100 indicates "extreme fatigue."
Pain Intensity While Coughing (VAS) | Baseline, 12 hours, 24 hours, and 48 hours post-intervention
  Pain experienced during coughing will be measured using a 100 mm Visual Analog Scale, where 0 represents "no pain" and 100 represents "worst possible pain."
Pain Intensity at Rest (VAS) | Baseline, 12 hours, 24 hours, and 48 hours post-intervention
  Participants will rate their resting pain intensity using a 100 mm Visual Analog Scale (VAS), where 0 is "no pain" and 100 is "worst pain imaginable."

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (de-identified) that underlie the results reported in this study will be made available upon reasonable request from qualified researchers, following publication. Data will be shared through institutional approval processes in accordance with ethical guidelines.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified individual participant data will be made available beginning 6 months after publication of the primary results and will remain available for up to 3 years upon request.
Access Criteria: Researchers may request access to the de-identified individual participant data (IPD) and supporting documents (e.g., protocol, SAP, ICF, analytic code) by submitting a written proposal that includes a clear research question and analysis plan. Requests should be sent to the Principal Investigator via institutional email. All requests will be reviewed by the research team and relevant ethics committee. If approved, data will be shared under a formal data use agreement. Data will be provided through a secure, password-protected digital platform.